CLINICAL TRIAL: NCT05199584
Title: A Phase 2, Multi-Center Study Evaluating the Safety and Efficacy of ENV-101 (Taladegib) in Patients With Advanced Solid Tumors Harboring PTCH1 Loss of Function Mutations
Brief Title: A Study Evaluating the Safety and Efficacy of ENV-101 (Taladegib) in Patients With Advanced Solid Tumors Harboring PTCH1 Loss of Function Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Endeavor Biomedicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENV-ONC-101
Record Dates: First submitted 2021-12-14; First posted 2022-01-20 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumors With PTCH1 Loss-of-function Mutations
Keywords: Patched-1; PTCH1; Hedgehog inhibitor; Smoothened inhibitor; Endeavor; NGS; Next Generation Sequencing; Head and Neck; Laryngeal; Hypopharyngeal; Nasal Cavity; Nasopharyngeal; Oral Cavity; Oropharyngeal; Throat; Salivary Gland; Lung; Lung Carcinoid; Breast; Skin; Basal; Squamous; Melanoma; Merkel Cell; Anal; Bile Duct; Colorectal; Esophagus; Gallbladder; Gastrointestinal; Liver; Pancreatic; Pancreatic Neuroendocrine Tumor; NET; Small Intestine; Stomach; Cervical; Endometrial; Ovarian; Penile; Prostate; Testicular; Uterine; Vaginal; Vulvar; Bone; Osteosarcoma; Rhabdomyosarcoma; Soft Tissue Sarcoma; Eye; Ocular Melanoma; Retinoblastoma; Brain; Spinal Cord; Neuroblastoma; Adrenal; Pituitary; Bladder; Kidney; Medulloblastoma; Glioma; Wilms; Precision Oncology; Mesothelioma
MeSH Terms: conditions — Laryngeal Diseases; Melanoma; Adenoma, Islet Cell; Osteosarcoma; Rhabdomyosarcoma; Sarcoma; Uveal Melanoma; Retinoblastoma; Neuroblastoma; Pituitary Diseases; Medulloblastoma; Glioma; Mesothelioma | interventions — LY2940680

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg ENV-101 (Experimental): ENV-101 (taladegib) tablets, 200 mg once-daily in 28-day cycles
  Interventions: Drug: ENV-101 (taladegib)
- 300 mg ENV-101 (Experimental): ENV-101 (taladegib) tablets, 300 mg once-daily in 28-day cycles
  Interventions: Drug: ENV-101 (taladegib)

INTERVENTIONS:
Drug: ENV-101 (taladegib) — tablets dosed once-daily

SUMMARY:
This study employs a 2-stage design that aims to evaluate the efficacy and safety of ENV- 101, a potent Hedgehog (Hh) pathway inhibitor, in patients with refractory advanced solid tumors characterized by loss of function (LOF) mutations in the Patched-1 (PTCH1) gene. Stage 1 of this study will enroll approximately 44 patients randomized between two dose levels. As appropriate, Stage 2 of the study will expand enrollment based on the results of Stage 1.

ELIGIBILITY:
Inclusion Criteria:

* Females or males greater than or equal to 18 years of age. If under 18 years of age, males must have a bone age of at least 17 years and females must have a bone age of at least 15 years. X-rays will be reviewed by a qualified physician (e.g. radiologist or endocrinologist) for eligibility for those under 18 years of age
* Has histologically or cytologically confirmed solid tumor that harbors a PTCH1 loss of function mutation, identified via genomic sequencing routinely performed at a CLIA certified laboratory
* Able to take medication orally
* Patients must be refractory to all standard of care therapy, or standard or curative therapy does not exist, or the patient has documented their refusal of standard of care therapies
* Patients willing to sign and have a full understanding of the informed consent form
* Life expectancy of ≥ 3 months

Exclusion Criteria:

* Concurrent administration of any anti-cancer therapies (e.g., chemotherapy, other targeted therapy) other than those administered in this study
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures. Patients with indwelling catheters are allowed
* Malignancies other than the primary tumor type within 5 years prior to study start, with the exception of those with a negligible risk of metastasis or death (e.g., expected 5-year Overall Survival > 90%) treated with expected curative outcome (e.g., in situ melanoma, basal or squamous cell skin cancer if completely excised, localized prostate cancer that is managed by surveillance, ductal carcinoma in situ treated surgically with curative intent are allowed)
* History of clinically significant autoimmune disease requiring prescription systemic therapy in the last two years prior to study start; patients with controlled hypothyroidism may be considered after evaluation by the Investigator.
* Presence of active infection at study start or confirmed active human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV)
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to study start, unstable arrhythmias, or unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician
* Refractory nausea and vomiting, malabsorption, external biliary shunt or significant bowel resection that would preclude adequate absorption of investigational product
* Major surgical procedure within 28 days prior to study start or anticipation of need for a major surgical procedure during the course of the study
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 28 days prior to study start
* Use of drugs that are known moderate or stronger CYP3A4 inhibitors or inducers within 12 days prior to study start
* Unresolved toxicity of ≥ CTCAE Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, platinum-induced neurotoxicity and endocrine disease or ailments that are stable)
* Males and females of reproductive potential who are sexually active and unwilling to use birth control for the duration of the study and for 3 months after their final study dose
* Females that are pregnant or nursing
* Females and males that are unwilling to refrain from blood or blood product donation for the duration of the study and for 30 days after their final study dose
* Males who are unwilling to refrain from sperm donation and females who are unwilling to refrain from egg donation for the duration of the study and for 3 months after their final study dose
* Patients with a history of a severe allergic reaction, anaphylactic reaction or known hypersensitivity to any component of ENV-101
* Patients who are immediate family members (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with a study investigative site or the study Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 6 months
  ORR is comprised of Complete Response (CR) and Partial Response (PR), measured by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1), as determined by an independent review (confirmed CR or PR will be defined as a repeat assessment performed no less than 28 days after the criteria for response is first met).

SECONDARY OUTCOMES:
Frequency of Adverse Events (AEs) | through study completion, an average of 6 months
Frequency of unacceptable toxicities | through study completion, an average of 6 months
  Unacceptable toxicities = non-hematologic AEs >= Grade 3 in severity, not including alopecia and fatigue.
ORR by Investigator | through study completion, an average of 6 months
  Best overall response of confirmed CR or PR as determined by the treating Investigator using RECIST 1.1.
Clinical Benefit Rate (CBR) | through study completion, an average of 6 months
  CBR = the proportion of patients who achieved CR, PR or stable disease as determined by the treating Investigator using RECIST 1.1.
Overall Survival (OS) | through study completion, an average of 6 months
  OS = Number of months from initiation of study medication to the date of death due to any cause or last follow up.
Duration of Response (DOR) | through study completion, an average of 6 months
  DOR = the number of months from the start of CR or PR, whichever response is recorded first and subsequently confirmed, to the first date that recurrent or progressive disease is documented or death.
Progression Free Survival (PFS) | through study completion, an average of 6 months
  PFS = number of months from initiation of study medication to the earlier of disease progression or death due to any cause or last follow up.
Change in Gli1 inhibition | From Baseline through study completion, an average of 6 months
  Percentage change in inhibition of Gli1, a marker for inhibition of the Hedgehog pathway, in skin biopsies.
Change in steady-state exposure to study medication | From Baseline through study completion, an average of 6 months
  Measurement of trough concentration of study medication in blood at Baseline and the end of each 28-day treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Paul Frohna, M.D., Ph.D., Study Director — Endeavor Biomedicines
Locations (16):
- United States (16):
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, Tampa, Florida
  - Research Site, Zion, Illinois
  - Research Site, Covington, Louisiana
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Fredericksburg, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No